CLINICAL TRIAL: NCT00446407
Title: The Effectiveness and Cost-effectiveness of a Collaborative Stepped Care Intervention for the Treatment of Common Mental Disorders in Primary Care Settings in Goa, India
Brief Title: Evaluating the Benefits and Affordability of a Program to Improve the Care of Common Mental Disorders in Primary Care
Acronym: MANAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); Sangath (Other); Voluntary Health Association of Goa, India (Other); Government of Goa, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MANAS
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2009-07

CONDITIONS: Depressive Disorders; Anxiety Disorders; Depression
Keywords: Depression; Primary Care; Developing Countries; Common mental disorders (depressive and anxiety disorders)
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collaborative Stepped Care (Experimental): Screening, Antidepressants, Psychosocial interventions (psychoeducation, IPT, adherence management) by Health Counselor, support and supervision by Psychiatrist.
  Interventions: Other: Collaborative Stepped Care Intervention
- Enhanced Usual Care (Active Comparator)
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Collaborative Stepped Care Intervention — Psychoeducation, interpersonal therapy, fluoxetine (20-40 mg/d), adherence management
  Arms: Collaborative Stepped Care
Other: Enhanced Usual Care — Screening plus Antidepressants based on practice guidelines
  Arms: Enhanced Usual Care

SUMMARY:
Depressive and anxiety disorders (termed as 'Common Mental Disorders') affect as many as one in four persons attending primary care; most patients do not receive effective treatments. Although the integration of mental health in primary care is accepted as the only feasible way of managing Common Mental Disorders in developing countries, there is no evidence demonstrating how this can be done in a manner which is effective and affordable. The hypothesis of this trial is that a Collaborative Stepped Care package will be both clinically and cost-effective for the treatment of Common Mental Disorders in primary care.

DETAILED DESCRIPTION:
The goal of the research is to evaluate the clinical and cost-effectiveness of a Collaborative Stepped Care intervention for the treatment of Common Mental Disorders (CMD) in primary care in Goa, India.

The Collaborative Stepped Care intervention will be compared with Enhanced Usual care in a cluster randomized controlled trial in 24 primary care facilities; the first phase of the trial will be located in 12 government run Primary Health Centres, while the second phase will be located in 12 private family physician/general practice facilities. Approximately 2400 participants who screen positive on a screening questionnaire for CMD will be recruited from the 24 facilities (a harmonic mean of 100 per cluster per arm) of whom 2/3 will be ICD10 cases confirmed by a diagnostic interview (the Revised Clinical Interview Schedule). Follow-up interviews at home will be conducted by an independent team at 2, 6 and 12 months post recruitment. Allowing for 25% attrition during follow-up gives 650 patients in each arm with a confirmed CMD, or a total of 960 in each arm, contributing to analyses of the primary outcomes (see below).

The Collaborative Stepped Care intervention is a complex intervention comprising the following components: screening for detection of cases; psycho-education; antidepressants; inter-personal therapy; yoga; specialist supervision & adherence management. The method of delivery will be based on the stepped-care model which provides treatments according to the patients' needs and incorporates strategies to overcome challenges to the integration of mental health in primary care in developing countries. This will be compared with Enhanced Usual Care which will comprise screening for detection of cases, provision of the diagnosis to the doctor, and making antidepressants available in the facility-all these components will be available in the Collaborative Stepped care facilities as well. The intervention will be delivered by two new, full-time, primary care human resources-the Health Assistant (in both arms) who will screen adult attenders; and in the Collaborative Stepped Care arms, the Health Counselor-who has been trained over 3 months, and a part-time Psychiatrist supporting the primary care team.

The primary analyses will be intention-to-treat, regardless of adherence to the intervention, and will be based on outcomes measured at 6 months. All analyses will take into account any within-facility clustering resulting from the cluster randomized design, and will include adjustment for any of the a-priori defined confounding factors for which randomization did not achieve balance between the two arms at baseline.

The primary research question being answered and the analysis outputs are:

* Does the Collaborative Stepped Care Intervention have an effect on the outcome of Definite Cases? Prevalence of CMD in the two arms amongst participants who had an International Classification of Diseases, tenth edition (ICD10) CMD at baseline
* Does the Collaborative Stepped Care Intervention have an effect on the burden of CMD amongst patients who are Possible Cases? Prevalence of CMD in the two arms in all screen-positive participants
* Does the Collaborative Stepped Care Intervention have an effect on the outcome of Depression Cases? Prevalence of CMD in the two arms amongst participants who had an ICD10 Depression at baseline
* Does the Collaborative Stepped Care Intervention have an effect on the incidence of ICD10 CMD amongst Sub-threshold Cases? Prevalence of CMD in the two arms in screen-positive participants who did not have an ICD10 CMD diagnosis at baseline.

Secondary analyses will include:

* Comparison of prevalences listed above at 2 months (as a measure of speed of recovery) and at 12 months (sustainability of effectiveness).
* Repeated measures analysis of CMD prevalence at 2, 6 and 12 months, to assess effect of the intervention over the whole 12 month follow-up period.
* Comparisons of Revised Clinical Interview Schedule (CISR) and General Health Questionnaire (GHQ) scores, and World Health Organisation Disability Assessment Schedule (WHO-DAS) scores as continuous outcomes (i) at each endpoint; and (ii) using repeated measures analyses combining information from the three endpoints.
* Interaction of gender, education and co-morbidity with intervention effects
* Interaction of facility type (private/public) with intervention effects.
* Interaction of baseline illness attribution (somatic/psychosocial) with intervention effects.
* Interaction of baseline severity of CISR scores with intervention effects
* Comparison of adverse events between the two arms at 2, 6 and 12 months.
* Per-protocol analysis:

  * Adherence with minimum intervention (at least one meeting with the Health Counselor in the Collaborative Stepped Care arm)
  * Adherence with optimal intervention-completion of intervention-i.e. discharge by the Health Counselor; or minimum therapeutic dose of either antidepressant (90% adherence over 90 days) or Interpersonal Psychotherapy (IPT) (6 sessions over 4 months).
  * Dose response relationship with levels of adherence

For the economic analysis, health care costs and other patient- or family-borne costs will be computed and compared at 2, 6 and 12 months, and subsequently related to changes in health outcome: both the primary outcome measure of depression status and also Quality Adjusted Life Years [QALYs]. In the event that dominance is not shown, i.e. the intervention is more effective but the costs are also more than the usual care group, incremental cost-effectiveness ratios will be computed, together with their confidence intervals (using bootstrapping techniques to overcome expected skewness of cost data). Cost-effectiveness acceptability curves will also be derived in order to show the probability of any cost-effective advantages for the component interventions at a range of 'willingness to pay' threshold levels.

We will also carry out a nested qualitative evaluation with the objective is to assess the participants' perceptions of the quality of the care they received, their satisfaction with this care, the reasons why they did/did not take full advantage of the intervention offered, and the impact of their health problems on their daily lives, economic productivity and lives of family members. We will also explore their experience of being a trial participant (in particular, the experience of the informed consent procedure; reasons for participation; their understanding of randomization). Two in-depth interviews will be conducted with at least 96 participants, the first about 1 month after enrolment and the second interview about 6 months later. A second group of in-depth interviews will be carried out with members of the intervention team about the process of the intervention, its successes and limitations (on quality of care, on the PHC's overall function) and how future programs may address these. We aim to interview at least one doctor from each facility and one Health Counselor from each PHC (i.e. total of 24). Two in-depth interviews will be conducted with each staff member, the first about 2 months after the initiation of the program. The second interview will be conducted between 6 and 12 month after the initiation of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18;
* Suffering from a Common Mental Disorder (as defined by an a priori cut-off score on the 12 item General Health Questionnaire)
* Resident in the state (Goa) for the subsequent 12 months
* Not requiring urgent medical/surgical attention (e.g hospital admission)

Exclusion Criteria:

* Suffering from a cognitive or sensory impairment which makes participation in the evaluation difficult
* Not speaking Konkani, Marathi, Hindi or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2796 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Recovery from Common Mental Disorder (defined by ICD10) | 6 months

SECONDARY OUTCOMES:
Case of CMD among all screen-positive participants at 2, 6 and 12 months | 2, 6 and 12 months
Case of CMD among all sub-threshold cases | at 2, 6 and 12 months
Recovery from CMD (defined by ICD10) among the subgroup with ICD-10 Depression at baseline | at 2, 6 and 12 months
Psychological morbidity (mean scores) | at 2, 6 and 12 months
Disability levels | at 2, 6 and 12 months
Costs of illness | 2, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Sangath, Porvorim, Goa, India

REFERENCES:
- [Derived] Pillai A, Keyes KM, Susser E. Antidepressant prescriptions and adherence in primary care in India: Insights from a cluster randomized control trial. PLoS One. 2021 Mar 19;16(3):e0248641. doi: 10.1371/journal.pone.0248641. eCollection 2021. PMID 33739982
- [Derived] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Lay health worker led intervention for depressive and anxiety disorders in India: impact on clinical and disability outcomes over 12 months. Br J Psychiatry. 2011 Dec;199(6):459-66. doi: 10.1192/bjp.bp.111.092155. PMID 22130747
- [Derived] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, De Silva MJ, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Effectiveness of an intervention led by lay health counsellors for depressive and anxiety disorders in primary care in Goa, India (MANAS): a cluster randomised controlled trial. Lancet. 2010 Dec 18;376(9758):2086-95. doi: 10.1016/S0140-6736(10)61508-5. Epub 2010 Dec 13. PMID 21159375
- [Derived] Patel VH, Kirkwood BR, Pednekar S, Araya R, King M, Chisholm D, Simon G, Weiss H. Improving the outcomes of primary care attenders with common mental disorders in developing countries: a cluster randomized controlled trial of a collaborative stepped care intervention in Goa, India. Trials. 2008 Jan 25;9:4. doi: 10.1186/1745-6215-9-4. PMID 18221516
- See also: Link to primary UK academic institution leading the trial — http://www.lshtm.ac.uk
- See also: Link to primary Indian organization leading the trial — http://www.sangath.com